CLINICAL TRIAL: NCT06554379
Title: Investigation of the Effect of Periodontal Health on Smile Parameters: a Cross-Sectional
Brief Title: The Effect of Periodontal Health on Smile
Acronym: EPHS
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Tuğba ŞAHİN, Assistant professor, Abant Izzet Baysal University
Other Study IDs: AIBU-DH-TS
Record Dates: First submitted 2024-08-11; First posted 2024-08-15 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Smiling; Gingival Diseases
Keywords: gingivitis; periodontal health; smile
MeSH Terms: conditions — Smiling; Gingival Diseases; Gingivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Periodontal health: It includes gingival healthy individuals without any periodontal disease.
  Interventions: Other: Periodontal health and gingivitis
- Gingivitis: It includes individuals with gingivitis.
  Interventions: Other: Periodontal health and gingivitis

INTERVENTIONS:
Other: Periodontal health and gingivitis — The presence or absence of periodontal disease in the gingiva was determined.

SUMMARY:
Anamnesis was taken from 108 patients aged 18-33 who applied to the clinic and met the inclusion criteria. Photographs of the patients' smiles were taken without any measurement. Plaque , gingival index , bleeding on probing, pocket depth measurements, clinical attachment, and gingival recession levels were measured, respectively. Patients were divided into two groups: peri-implant health and gingivitis. Gingival thickness and keratinized gingival width were also measured. In addition, the smile aesthetic index, style, type, and stage were also determined using the smile classification system. Gingival visibility was measured in mm from the photographs taken.

ELIGIBILITY:
Inclusion Criteria:

* No systemic disease

Exclusion Criteria:

* Active smoking,
* Ongoing or past orthodontic treatment,
* Pregnancy,
* Nursing,
* Individuals who have drug-induced gingival hyperplasia, hereditary gingival fibromatosis, permanent or removable prostheses in the upper front area, or missing teeth in the front region

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 108 systemically healthy individuals between 13 and 33 years of age
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Keratinized gingival thickness | Baseline
  Keratinized gingival thickness refers to the vertical measurement of the gingival tissue that extends from the free gingival margin to the mucogingival junction, characterized by a keratinized epithelial layer which provides enhanced protection and stability to the underlying periodontal structures.
Keratinized gingival width | Baseline
  Keratinized gingival width refers to the horizontal dimension of the gingival tissue that is keratinized, measured from the free gingival margin to the mucogingival junction.
Gingival display | Baseline
  The gingival displays were measured by measuring the distances from the zenith points to the vermilion border
Smile esthetic index | Baseline
  . The aforementioned factors were assigned a number (0 or 1) depending on their presence or absence, and the total of the assigned numbers indicates the subject's SEI (which ranges from 0 for very poor to 10 for very good)
Smile clasificatain system | Baseline
  Smile style (Commissura smile, sharp smile, and complex smile), stage (Stage I, Stage II, Stage III, and Stage IV), and type (Type 1, Type 2, Type 3, and Type 4) were analyzed with the smile classification system
Gingival phenotype | Baseline
  The visible end of the periodontal probe in the sulcus represents a thin gingival phenotype, while the invisible end corresponds to a thick gingival phenotype

SECONDARY OUTCOMES:
Plaque index | Baseline
  The plaque index assesses the amount of dental plaque visible on the vestibular and lingual surfaces of all teeth
Gingival index | Baseline
  This measurement is based on the presence or absence of bleeding on gentle probing
Bleeding on probing | Baseline
  Bleeding, leading sign of inflammation inside the connective tissue, is a critical factor for pocket depth measurements, and with other variable factors prevents making reproducible measurements.
Periodontal pocket depth | Baseline
  A pathologically deepened gingival sulcus around a tooth at the gingival margin.
Clinical attachment level | Baseline
  CAL is calculated by subtracting the gingival margin level from the probing depth.
Gingival recession depth | Baseline
  Gingival recession is the apical migration of the gingival margin away from the cemento-enamel junction (CEJ), resulting in the exposure of the root surface of a tooth.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Bolu, Turkey (Türkiye)